CLINICAL TRIAL: NCT03989024
Title: Pulsatile Gonadotropin-releasing Hormone for Infertility in Non-obese Patients With Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18411968700
Record Dates: First submitted 2019-05-30; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Polycystic Ovary Syndrome; Infertility; Ovulation Disorder
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Gonadotropin-Releasing Hormone; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pulsatile Gonadotropin-releasing Hormone (Experimental): Drug: Gonadorelin. Use Gonadorelin for 3 months to treat PCOS. The pulse was administered with a hormone pump, once every 90 min, and 10ug per pulse.
  Interventions: Drug: Gonadorelin
- Clomiphene (Experimental): Use Clomiphene for 3 months to treat PCOS
  Interventions: Drug: Clomiphene

INTERVENTIONS:
Drug: Gonadorelin — Drug: Gonadotropin-releasing Hormone. Generic name: Gonadorelin. Dosage form: 600ug. Dosage: 10ug/puls. Frequency: every 90 min. Duration: 3 months
  Arms: Pulsatile Gonadotropin-releasing Hormone
Drug: Clomiphene — Drug: Clomiphene. Generic name: Clomiphene. Dosage form: 50mg. Dosage: 50mg. Frequency: once a day. Duration: 3 months
  Arms: Clomiphene

SUMMARY:
Polycystic ovary syndrome (PCOS) patients are often accompanied by infertility. Non-obese PCOS infertility is more difficult to treat than obese PCOS. The study included non-obese PCOS patients who had not recovered from regular menstruation after six months of metformin treatment. Half of the patients were treated with clomiphene for ovulation induction and half with GnRH pulse therapy.

DETAILED DESCRIPTION:
To investigate whether GnRH pulse therapy of non-obese PCOS women can improve ovulation rate.The investigators plan to recruit non-obese PCOS women with abnormal GnRH pulse mode not effective of metformin treatment at childbearing age. By using GnRH pulse therapy and Clomiphene therapy. the investigators will intervent the participants for 3 months and to compare outcome in each group.

ELIGIBILITY:
Inclusion Criteria:

1. PCOS of childbearing age (24-45 years old);
2. non-obesity;
3. After 6 months of metformin (at least 1000-1500 mg/d) intervention, the normal menstrual cycle was still not restored.
4. No drug intervention except metformin was used in last 3 monthes:
5. There is a pregnancy plan within 1 years.
6. The pregnancy test was negative.
7. Heart and liver function is normal, thyroid function is normal, adrenal function is normal.
8. The GnRH stimulation test confirmed that the pituitary and ovarian reserve function was good.
9. Chromosome examination is normal.
10. Did not take part in other clinical trials.

Exclusion Criteria:

1. PCOS was not diagnosed.
2. Severe liver and kidney dysfunction (ALT is 2.5 times greater than normal upper limit, or Cr > 132 umol/l, or eGFR < 60 mL/min/1.73 m2), thyroid dysfunction, adrenal dysfunction, psychosis, severe infection, severe anemia, neutropenia;
3. Other serious organic heart diseases, such as congenital heart disease, rheumatic heart disease, hypertrophic or dilated cardiomyopathy, NYHA cardiac function grade (> III);
4. Kallmann syndrome, secondary hypogonadotropic hypogonadism, acquired central nervous system diseases, infertility caused by hypothalamic amenorrhea and other secondary infertility;
5. Has a history of abuse of active substances, including alcohol and a history of alcohol related diseases in the past 2 years.
6. Previous history of central nervous system and gonad-related surgery, or other central nervous system and gonad-related surgery (such as central nervous system tumor resection, ovarian chocolate cyst resection) within one year, or other non-central nervous system and gonad surgery within six months;
7. In the past five years, there have been organ system tumors (except for local cutaneous basal cell carcinomas) that have been treated or not treated, regardless of whether there is evidence of local recurrence or metastasis;
8. Hypoglycemic drugs, contraceptives (Dain, Marvelon), ovulation-promoting drugs (clomiphene, letrozole), emergency contraceptives and sex hormone drugs have been or are being used to adjust menstrual cycle and promote ovulation except metformin.
9. Pregnancy;
10. GnRH stimulation test confirmed pituitary and ovarian reserve dysfunction.
11. Abnormal chromosome detection.
12. Patients who are allergic to drugs with similar chemical structure.

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ovulation recovery (according to basal body temperature, progesterone levels on cycle day 21, or ultrasonography) | up to 12 weeks
  Number of participants with ovulation recovery (according to basal body temperature, progesterone levels on cycle day 21, or ultrasonography) after use of drugs

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 12 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. Evaluation of efficacy and safety of short-term GnRH pulse therapy for non obese PCOS

CONTACTS AND LOCATIONS:
Overall Officials: TAO TAO, DM, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No